CLINICAL TRIAL: NCT06735781
Title: Short-term Clinical Outcomes of Patients With Resectable Non-Small Cell Lung Cancer Receiving Nivolumab Plus Chemotherapy as Neoadjuvant Therapy in France
Brief Title: Clinical Outcomes of Patients With Resectable Non-Small Cell Lung Cancer Receiving Neoadjuvant Nivolumab Plus Chemotherapy in France
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-1512
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
Keywords: Non-small cell lung cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neoadjuvant nivolumab plus chemotherapy treatment
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — As prescribed by the treating clinician

SUMMARY:
The purpose of this study is to evaluate real-world effectiveness of neoadjuvant nivolumab plus chemotherapy in France.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of resectable non-small cell lung cancer (NSCLC)
* Being 18 years or above at the time of their NSCLC diagnosis
* Having initiated a neoadjuvant treatment with nivolumab and chemotherapy outside a clinical trial
* Being indexed in the site database
* Being followed at the site for at least 5 months, except for patients with a record of death

Exclusion Criteria:

• Having any primary tumor other than NSCLC on or before the date of NSCLC diagnosis that required a treatment ending less than 12-months before the nivolumab plus chemotherapy neoadjuvant treatment

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will include adults that have been diagnosed with resectable non-small cell lung cancer who initiated nivolumab plus chemotherapy as neoadjuvant therapy outside of clinical trial setting in France
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2024-09-05 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Rate of pathological complete response on date of surgery | Up to 31 months (until loss of follow-up, death, or end of study observation period)

SECONDARY OUTCOMES:
Study population baseline demographics | Baseline
Study population baseline clinical characteristics | Baseline
Surgery rate | Up to 31 months (until loss of follow-up, death, or end of study observation period)
Time from diagnosis to start of neoadjuvant treatment | Up to 31 months (until loss of follow-up, death, or end of study observation period)
Average dose of nivolumab infusions | Up to 31 months (until loss of follow-up, death, or end of study observation period)
Frequency of nivolumab infusions | Up to 31 months (until loss of follow-up, death, or end of study observation period)
Duration of nivolumab treatment | Up to 31 months (until loss of follow-up, death, or end of study observation period)
Type of chemotherapy received in combination with nivolumab treatment as neoadjuvant treatment | Up to 31 months (until loss of follow-up, death, or end of study observation period)
Infusion setting (hospital or at home) | Up to 31 months (until loss of follow-up, death, or end of study observation period)
Survival status | at 3, 6, 9, 12, 18, and 24 months (or until loss of follow-up, death, or end of study observation period (31 months))
Subsequent treatments received after nivolumab treatment | Up to 31 months (until loss of follow-up, death, or end of study observation period)
Disease progression/relapse status | At 3, 6, 9, 12, 18, and 24 months (or until loss of follow-up, death, or end of study observation period (31 months))
Rate of major pathological response | Up to 31 months (until loss of follow-up, death, or end of study observation period)
Adverse events | Up to 31 months (until loss of follow-up, death, or end of study observation period)
Time to surgery from initial diagnosis | Up to 31 months (until loss of follow-up, death, or end of study observation period)
Time to surgery from the first dose of neoadjuvant therapy | Up to 31 months (until loss of follow-up, death, or end of study observation period)
Time to surgery from the last dose of neoadjuvant therapy | Up to 31 months (until loss of follow-up, death, or end of study observation period)
Surgery type | Up to 31 months (until loss of follow-up, death, or end of study observation period)
Duration of surgery | Up to 31 months (until loss of follow-up, death, or end of study observation period)
Extent of surgical resection | Up to 31 months (until loss of follow-up, death, or end of study observation period)
Rate of lymph node resection | Up to 31 months (until loss of follow-up, death, or end of study observation period)
Type of surgery complications | Up to 31 months (until loss of follow-up, death, or end of study observation period)
Length of hospital stay | Up to 31 months (until loss of follow-up, death, or end of study observation period)
Reasons for not having surgery as indicated by the multi-disciplinary tumor board | Up to 31 months (until loss of follow-up, death, or end of study observation period)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (7):
- France (7):
  - Centre François Baclesse, Caen
  - Centre Léon Bérard, Lyon
  - Hospices Civils de Lyon, Lyon
  - Hôpital Robert Schuman, Metz
  - Institut du Cancer de Montpellier, Montpellier
  - Institute Curie, Paris
  - Hôpital d'Instruction des Armées Saint Anne, Toulon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts